CLINICAL TRIAL: NCT04887116
Title: Piloting Virtual Reality Environments to Treat PTSD in Healthcare Workers
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-04021926
Record Dates: First submitted 2021-05-13; First posted 2021-05-14 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; Virtual reality; VR; Healthcare workers; COVID-19; Pandemic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; COVID-19 | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Exposure Therapy (Experimental): Virtual Reality Exposure Therapy
  Interventions: Behavioral: Virtual Reality Exposure Therapy

INTERVENTIONS:
Behavioral: Virtual Reality Exposure Therapy — Ten ninety minute sessions of Virtual Reality Exposure Therapy twice a week for five weeks, either remotely or in person.

SUMMARY:
Healthcare workers and COVID-19 patients may experience psychological distress consequent to the pandemic, and are at particularly elevated risk for experiencing posttraumatic stress disorder (PTSD), based on evidence from previous infectious disease outbreaks. The best-validated treatment for PTSD is exposure therapy. Exposure therapy help patients suffering from PTSD to revisit and overcome their traumatic experiences. Including virtual reality in exposure therapy has a long history in treating PTSD; and has been used to treat military veterans and first-responders following 9/11. The investigators are developing and testing a virtual environment to treat PTSD including sub threshold PTSD symptoms in HCWs who experience occupational related trauma (e.g., working with COVID-19 patients) and COVID-19 patients. An independent evaluator will assess symptoms of PTSD and other psychopathology, using structured clinical interviews and self-report measures with well-established psychometric properties, at baseline, halfway through treatment, after completion of treatment, and at three-months post-treatment. Participants will complete ten ninety minute sessions (in-person or remotely), twice a week for five weeks aimed at mitigating their symptoms of PTSD. Remote participants will receive VR headsets after the baseline assessment and will keep them for the duration of the study. The pilot study will aim to demonstrate the feasibility and the tolerability of the virtual reality intervention in these populations.

ELIGIBILITY:
Inclusion Criteria:

* A COVID-19 patient or any healthcare worker providing medical care or support who experiences occupational-related trauma
* English-speaking
* Age ≥18
* Medically stable
* Diagnosed with PTSD or sub threshold PTSD
* Ability to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments
* Stable on psychotropic medication for the prior 60 days

Exclusion Criteria:

* Current significant unstable medical illness such that the participant could not attend sessions regularly or complete assessments
* Patients who in the investigator's judgment pose a current homicidal, suicidal or other risk
* Lifetime or Current diagnosis of schizophrenia or other psychotic disorder
* Participation in a clinical trial or concurrent evidence-based treatment for psychiatric conditions or PTSD during the previous 3 months
* History of motion sickness or seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in Clinician Administered PTSD Score (CAPS-V) | Baseline to approximately five weeks
  Change in Clinician-Administered PTSD Scale for DSM-5 (CAPS-V) Score. Total Scores range from 0-80. Higher scores indicate greater symptom severity.
Feasibility Indicator: Recruitment | Baseline
  Feasibility assessment will include recruitment defined as number of individuals interested in the intervention.
Feasibility Indicator: Enrollment | Baseline
  Feasibility assessment will include enrollment defined as number of participants signing the informed consent form.
Feasibility Indicator: Retention | Post-Treatment Assessment at approximately 5 weeks
  Feasibility assessment will include retention defined as the number of participants completing the full intervention.
Acceptability Indicator: Satisfaction | Post-Treatment Assessment at approximately 5 weeks
  Acceptability and treatment satisfaction will be rated with a Likert scale.

SECONDARY OUTCOMES:
Change in Anxiety Symptoms measured by the Generalized Anxiety Disorder 7-Item Scale | Baseline to approximately five weeks
  Scored between 0-21:
  Cut offs:
  0-4 = None 5-9 = Mild anxiety 10-14 = Moderate anxiety 15-21 = Severe anxiety Higher scores indicate greater symptom severity.
Change in Depressive Symptoms measured by the Quick Inventory of Depressive Symptomatology | Baseline to approximately five weeks
  16-item self-report measure. Scored between 0-27. Higher scores indicate greater symptom severity.
Change in score on the Insomnia Sleep Index | Baseline to approximately five weeks
  7 item self-report measure. Total scores range from 0-28, with higher scores indicating higher insomnia severity.
Change in score on the PTSD Checklist for DSM-5 (PCL-5) | Baseline to approximately five weeks
  The well-validated PCL-5 will assess self-reported PTSD symptom severity. Scores range from 0-80. Higher scores indicate greater symptom severity.
Change in Score on the Occupational Stress Inventory Revised (OSI-R) | Baseline to approximately five weeks
  The scale is comprised of 140 items total. The measure is comprised of 14 different scales and respondents indicate on a 5-point scale the frequency of a stress-related event.
Change in score on the Modified Moral Injury Events Scale | Baseline to approximately five weeks
  11 item self-report measure that measures moral injury. Statements related to distress or feelings of betrayal related to potentially morally injurious events are rated on a 6 point scale ranging from 1 (strongly agree) to 6 (strongly disagree).
  Score range is 11-66, with higher scores reflecting greater moral injury.
Change in score on the Sheehan Disability Scale (SDS) | Baseline to approximately five weeks
  10 point visual analog scale to rate the extent to which work/school, social life and home life or family responsibilities are impaired by his or her symptoms. The 3 items can be summed into a single dimensional measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired).
Change in score on the Social Adjustment Scale (SAS) | Baseline to approximately five weeks
  Subjects rate their own social functioning over times on a 5-point scale on items covering work for pay, housework, extended family, parenting, marital status, social activity and leisure, family unit and student status (sub-scales). Mean values of all the sub-scales are used, with a range from 0-5. Higher score = worse outcome.
Change in score on the Moral Distress Scale | Baseline to approximately five weeks
  21 item self-report measure measuring moral distress (the emotional state that arises from a situation when an individual feels that the ethically correct action to take is different from what he/she is tasked with doing). Score range is 0-336. Higher scores indicate greater moral distress.
Change in score on the Quality of Life Inventory | Baseline to approximately five weeks
  The assessment yields an overall score and profile in 16 areas of life; health, self-esteem, goals and values, money, work, play, learning, creativity, helping, love, friends, children, relatives, home, neighbourhood, and community. Higher scores indicate higher level of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: JoAnn Difede, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No